CLINICAL TRIAL: NCT06448468
Title: Analysis of Ocular Surface Microbiota in Dry Eye Patients After Femtosecond Laser-assisted In-situ Keratomileusis (FS-LASIK)
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Yifeng Yu, Deputy chief physician of Ophthalmology center of the Second Affiliated Hospital of Nanchang University, Second Affiliated Hospital of Nanchang University
Other Study IDs: [2024] No. (34).
Record Dates: First submitted 2024-05-27; First posted 2024-06-07 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Refractive Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dry group
- Non dry eye group

SUMMARY:
By using 16S rRNA sequencing technology to analyze the changes in ocular surface microbiota before and after surgery, as well as the impact of changes in ocular surface microbiota on FS-LASIK induced DES, new treatment ideas are provided for corneal FS-LASIK induced DES patients, and the incidence of FS-LASIK related DES is reduced.

DETAILED DESCRIPTION:
This study aims to include 160 postoperative patients, who will be divided into a dry eye group and a normal group based on postoperative dry eye examination. Microbial samples of the patient's conjunctival sac will be collected, and changes in the ocular surface microbiota before and after surgery will be analyzed using 16S rRNA sequencing technology. The impact of changes in the ocular surface microbiota on FS-LASIK induced DES will also be analyzed, providing new treatment ideas for FS-LASIK induced DES patients and reducing the incidence of FS-LASIK related DES.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Stable refractive index (refractive index change less than 0.5D in the past 2 years);
3. The best corrected far vision (CDVA) is 1.0 or better;
4. Postoperative dry eye patients need to meet the following criteria: Patient's Eye Surface Disease Index (OSDI) ≥ 13 and two of the following three criteria are met: Tear film rupture time (BUT) ≤ 10S Schirmer I test (mm/5min) ≤ 10mm, corneal fluorescein sodium staining exceeding 5 spots;

Exclusion Criteria:

1. History of eye trauma or surgery;
2. Suspected keratoconus;
3. Previously suffering from other eye diseases such as keratitis or edema, glaucoma, uveitis, retinal detachment, macular degeneration, cataracts, amblyopia, etc.;
4. Preoperative history of severe dry eye disease;
5. Patients with systemic diseases, such as hyperthyroidism or autoimmune diseases; Or severe mental disorders, such as anxiety and depression;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dry eye patients after FS-LASIK
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Sampling of conjunctival sac microbiota | Preoperative and Postoperative DAY 90
  Microbial diversity of conjunctival sac
Dry eye examination | Preoperative and Postoperative DAY 90
  Tear Film Break Up Time
Corneal nerve condition | Preoperative and Postoperative DAY 90
  corneal nerve fiber density
Dry eye examination | Preoperative and Postoperative DAY 90
  Schirmer Ⅰ test
Dry eye examination | Preoperative and Postoperative DAY 90
  ocular surface disease index
Corneal nerve condition | Preoperative and Postoperative DAY 90
  corneal nerve branch density
Corneal nerve condition | Preoperative and Postoperative DAY 90
  corneal nerve fibre length

CONTACTS AND LOCATIONS:
Locations (1):
- Yifeng Yu, Nanchang, Jiangxi, China